CLINICAL TRIAL: NCT04525586
Title: LncRNA and Predictive Model to Improve the Early Diagnosis of Childhood Asthma
Brief Title: lncRNA-based Nomogram to Assist Childhood Asthma Diagnosis
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: LLJ1.0
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Childhood Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- It's just an observational study, no interventions: children with recurrent wheezing

SUMMARY:
Asthma is the most common chronic disease in children, however, underdiagnosis of childhood asthma is an important issue in asthma management. The lack of reliable and objective diagnostic indicators requires the development of rapid and accurate strategies for the early diagnosis of childhood asthma. Recent studies have found a correlation between long-chain non-coding RNA (lncRNA) expression and childhood asthma, suggesting that lncRNA may be a potential biomarker for asthma diagnosis.

DETAILED DESCRIPTION:
The investigators envision exploring the early diagnosis of asthma by combining lncRNA with electronic medical records. In this project, the investigators will combine high-throughput sequencing, asthma case database, electronic medical record and informatics to investigate the feasibility of combining lncRNA with electronic medical record for asthma diagnostic model. The expected results will establish the foundation for the diagnosis and treatment of childhood asthma and open up new ideas.

ELIGIBILITY:
Inclusion Criteria:

children with recurrent wheezing

Exclusion Criteria:

1. diagnosis of other chronic respiratory disease (e.g. cystic fibrosis, bronchopulmonary dysplasia, etc)
2. immunodeficiency- acquired or congenital
3. neuromuscular disease
4. congenital heart disease

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with recurrent wheezing who apply to Department of Respiratory Medicine, Children's Hospital of Fudan University.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
rate of early diagnosis of childhood asthma | 24 months
  a diagnosis of transient wheeze or asthma was made by a pediatric pulmonologist. This classification was based on symptoms, use of asthma medication, and lung function features.

CONTACTS AND LOCATIONS:
Overall Officials: Liling Qian, PhD., Study Director — Children's Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No
The investigators do not currently have an individual participant data sharing plan. However, de-identified research data/documents may be shared in the future with other investigators who share similar research interests.
  Specimens and data will not be released without (1) PI written permission and (2) appropriate Institutional Review Board (IRB) approval. Data use and/or material transfer agreements will also be required as applicable to outside researchers.